CLINICAL TRIAL: NCT04262687
Title: Pembrolizumab in Combination With Xelox Bevacizumab in Patients With Microsatellite Stable Mestatic Colorectal Cancer and a High Immune Infiltrate : a Proof of Concept Study
Brief Title: Chemotherapy and Immunotherapy as Treatment for MSS Metastatic Colorectal Cancer With High Immune Infiltrate
Acronym: POCHI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1703 POCHI
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer Metastatic; High Immune Infiltrate; Microsatellite Stable
Keywords: immunotherapy; immune infiltrate; first line
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Bevacizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy + chemotherapy (Experimental): Xelox bevacizumab plus pembrolizumab every 3 weeks up until disease progression, unacceptable toxicity, refusal by the patient, withdrawal of consent, pregnancy or decision by the investigator.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Capecitabine — 2000 mg/m²/day, from day 1 to 14 of each cycle
Drug: Oxaliplatin — 130 mg/m² by IV infusion over 2 hours, on day 1 of each cycle
Drug: Bevacizumab — 7.5 mg/kg by IV infusion over 60 minutes, on day 1 of each cycle
Drug: Pembrolizumab — 200 mg by IV infusion over 30 minutes, on day 1 of each cycle

SUMMARY:
About 85% of cases of non-metastatic colorectal cancer (CRC) are related to chromosomal instability and have a proficient DNA Mismatch-Repair system (pMMR); which are also called CRC with microsatellite stability (MSS). Other CRC, i.e. 15%, are "microsatellite unstable" (MSI) with deficient DNA Mismatch-Repair system (dMMR). These latter are characterised by generation of many neo-antigens, which result in a high anti-tumour immune response and a high peri- and/or intra-tumour lymphocyte infiltration (TIL). Investigators recently showed, with a prospectively validated immune score, that 14% of localised MSS/pMMR CRC are also highly infiltrated by CD3+ lymphocytes. This same immune score has made it possible to measure high lymphocyte infiltration in hepatic metastases, in particular, in patients treated with XELOX/FOLFOX.

Pembrolizumab, an anti-PD1 monoclonal antibody (programmed death-1) is an immune checkpoint inhibitor (ICI) of PD1/PD-L1 axis, recently approved in many cancers. Anti-PD1 antibodies have recently been reported as being very effective in patients with dMMR metastatic CRC (mCRC). In the study by Le DT et al. pMMR mCRC did not seem to benefit from anti-PD1 antibodies. However, it is possible that 20% of pMMR mCRC with a high CD3+ infiltrate in the tumour may be a subgroup of pMMR mCRC sensitive to ICI, as is the case for dMMR mCRC. Lastly, immunogenic cell death induced by chemotherapy, such as oxaliplatin, can increase the efficacy of ICI.

The prognostic value of lymphocyte infiltrate has been demonstrated in CRC by several teams. However, no validated test is used in routine clinical practice. Previously, investigators described an automated and reproducible method for analysis of TIL and investigators validated it for clinical use. Automated tests evaluating TIL are performed on virtual slides and have showed that, out of 1,220 tumours tested, 20% were highly infiltrated by CD3+ T cells. Patients presenting with a pMMR CRC with a high immune infiltrate had a better progression-free survival (HR=0.70; p=0.02). An immunoscore® described by Galon et al. has also a high prognostic value in CRC and is based on CD3+ and CD8+ T cells infiltration in the center and periphery of the tumour. Finally, approximately 14% of tumours with a high immune infiltrate have been found in patients with metastatic CRC.

Investigators formulated the hypothesis that patients with a pMMR CRC with a high immune infiltrate can be sensitive to ICI . Therefore, blocks of resected primary tumour will be collected and analysed prospectively. For each patient, slides containing tumour tissue and adjacent non-tumour tissue will be analysed using two techniques : immunoscore® and TuLIS score.It consist in Immunohistochemistry with CD3 and CD8 staining. Slides will be scanned and analysed by image analysis as previously described . Tumours will then be classified as having a "high" or "low" immune response according to type of lymphocyte infiltrate, which is independent of pre-analytic conditions. Only patients with a high immune response will be eligible for the POCHI trial. Other biomarkers will be analysed like other immune populations or mutational load. If investigators identify an immune score which seems clinically relevant to predict sensitivity to ICI in pMMR mCRC, this will make it possible to plan a randomised phase III trial comparing chemotherapy and anti-angiogenic antibody versus chemotherapy and anti-angiogenic antibody plus pembrolizumab in patients with a pMMR mCRC with a high immune score and/or a hypermutated genotype.

Investigators choose PFS at 10 months as primary endpoint in POCHI trial because it is a surrogate marker of OS. Actually median PFS in first-line setting with a doublet plus a biological agent is range from 8 to 11 months in unresectable mCRC, corresponding to a PFS of 50% at 10 months. The alternative clinical hypothesis to obtain 70% of patients alive and without progression at 10 months is ambitious and currently not achieved with current chemotherapies plus a biological agent. Up until now there is no data concerning survivals outcomes of patients with a MSS mCRC with high immune infiltration score.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* MSS and pMMR metastatic colorectal adenocarcinoma (metachronous or synchronous metastases), histologically proven
* Patients who have had chemotherapy (neo-adjuvant or adjuvant) or radiotherapy (neo-adjuvant or adjuvant) for the treatment of primary tumor or metastatic resected disease R0 can be included if they have a recurrence more than 6 months after the end of this treatment.
* High immune response defined as the immune infiltration scores obtained on the primary tumour (resection of primary tumour containing at least 2 mm of tumour-free margin between the tumour and non-tumour area)
* Unresectable cancer with at least one measurable metastatic target according to RECIST v1.1 criteria
* WHO PS ≤ 1
* Life expectancy ≥ 3 months
* Adequate haematological function: neutrophils ≥ 1,500 /mm3, platelets ≥ 100,000/mm3, Hb > 9 g/dL
* Adequate liver function: AST/ALT ≤ 5xULN, total bilirubin ≤ 2xULN, alkaline phosphatase. ≤ 5xULN
* Creatinine clearance > 50 mL/min according to the MDRD formula
* Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour
* Patient who is a beneficiary of the social security system
* Information provided to patient and signature of the informed consent form

Exclusion Criteria:

* Active infection requiring intravenous antibiotics at day 1 of cycle 1
* Active or untreated central nervous system metastases
* Another concomitant cancer or history of cancer during the last 5 years, except for carcinoma in situ of the uterine cervix or a basal cell or squamous cell skin carcinoma or any other carcinoma in situ considered as cured
* Previous bone marrow allogenic stem cell transplantation or previous organ transplantation
* History of idiopathic pulmonary fibrosis, medicinal product-related pneumonia or proof of active pneumonia or pneumonitis on a chest CT-scan prior to therapy
* HIV infection, active hepatitis B or C infection, active tuberculosis
* Colorectal cancer with microsatellite instability (dMMR and/or MSI)
* Patient eligible for curative treatment (resection and/or thermal ablation according to the opinion of the local multidisciplinary tumour meeting board)
* Patient with only primary tumour biopsies available or only a sample of a metastasis (no surgical resection of the primary tumour)
* Previous treatment with anti-PD1 or anti-PDL1 or another immunotherapy
* An auto-immune disease which may worsen during treatment with an immune-stimulating agent (patients with type I diabetes, vitiligo, psoriasis, hypo or hyperthyroidism not requiring immunosuppressant therapy are eligible)
* Long-term immunosuppressant therapy (patients requiring corticosteroid therapy are eligible if administration at a dose ≤ 10 mg prednisone equivalent dose per day, administration of steroids by a route of administration resulting in minimal systemic exposure (cutaneous, rectal, ocular or inhalation) is authorised)
* Known severe hypersensitivity to monoclonal antibodies, to one of the medicinal products used or to one of the excipients in the products used or a history of anaphylactic shock or of uncontrolled asthma
* Vaccinations (live vaccine) within 30 days prior to start of treatment
* Dihydropyrimidine Dehydrogenase (DPD) deficiency defined by uracilemy level ≥ 16 ng/mL
* QT/QTc interval > 450 msec in men and > 470 msec in women
* One of the following disorders during the 6 months prior to inclusion: myocardial infarction, unstable/severe angina pectoris, coronary artery bypass grafting, NYHA class II, III or IV congestive heart failure, stroke or transient ischaemic attack
* All uncontrolled progressive disorders during the last 6 months: hepatic insufficiency, renal insufficiency, respiratory insufficiency, arterial hypertension
* History of an inflammatory digestive disease, obstruction or sub-obstruction not resolved with symptomatic treatment
* Peptic ulcer disease not healed before the treatment
* Not controlled HTA
* Patient already enrolled in another therapeutic trial with an ongoing investigational drug or whose treatment ended less than 4 weeks before inclusion
* Absence of effective contraception in patients (male and/or female patients) of childbearing potential, a pregnant or breastfeeding woman, women of childbearing potential and who have not had a pregnancy test
* Impossibility to submit to medical follow-up of the trial due to geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The rate of patients alive and without progression at 10 months after inclusion | 10 months after inclusion
  Progression is evaluated by CT scan, according to RECIST criteria (version 1.1) definition by the investigator. Death was also considered as an event (all causes). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed during the study (NADIR), or a measurable increase in a non-target lesion, or the appearance of new lesions

SECONDARY OUTCOMES:
Overall survival | Up to 2 years after the end of the treatment
  Overall survival is defined as the time from the date of the patient's inclusion to the patient's death (all causes). For alive patients the date of the latest news is taken into account
Histological response in case of secondary resection | Up to 2 years after the end of the treatment
  Response evaluated according to the TRG (Rubbia-Brandt L et al. Annals Oncol 2007), for patients who underwent a secondary resection

CONTACTS AND LOCATIONS:
Overall Officials: David TOUGERON, MD,PHD, Principal Investigator — CHU Poitiers
Locations (88):
- France (88):
  - Ch - Centre Hospitalier D'Abbeville, Abbeville
  - Chu - Hôpital Sud, Amiens
  - Privé - Clinique de L'Europe, Amiens
  - Privé - Ico - Site Paul Papin, Angers
  - Privé - Hôpital Privé Pays de Savoie, Annemasse
  - Privé - Hôpital Privé D'Antony, Antony
  - Ch - Hôpital Henri Duffaut, Avignon
  - Prive - Institut Du Cancer Avignon Provence, Avignon
  - Ch - Centre Hospitalier de La Côte Basque, Bayonne
  - Privé - Clinique Capio Balharra, Bayonne
  - Ch - Centre Hospitalier de Beauvais, Beauvais
  - Chu - Hôpital Jean Minjoz, Besançon
  - Ch - Centre Hospitalier de Béziers, Béziers
  - Privé - Cac - Clinique Bergonié, Bordeaux
  - Privé - Polyclinique Bordeaux Nord, Bordeaux
  - Privé - Clinique Tivoli, Bordeaux
  - Chu - Hôpital Ambroise Paré - Service Anatomie Pathologique, Boulogne
  - Ch - Hôpital Duchenne, Boulogne-sur-Mer
  - Chu - Hôpital Morvan - Institut de Cancérologie, Brest
  - Privé - Clinique Pasteur Lanroze Cfro, Brest
  - Privé - Centre Maurice Tubiana, Caen
  - Privé - Cac - Centre Francois Baclesse, Caen
  - Prive - Polyclinique Du Parc Caen, Caen
  - Privé - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Privé - Médipole de Savoie, Challes-les-Eaux
  - Privé - Hôpital Privé Paul D'Egine, Champigny-sur-Marne
  - Ch - Centre Hospitalier de Cholet, Cholet
  - Chu - Hôpital Estaing, Clermont-Ferrand
  - Ch - Hôpitaux Civils de Colmar, Colmar
  - Privé - Clinique Saint Come, Compiègne
  - Privé - Clinique de Flandre, Coudekerque-Branche
  - Ch - Ghpso - Site de Creil, Creil
  - Chu - Hôpital Henri Mondor, Créteil
  - Ch - Chic de Créteil, Créteil
  - Chu - Hôpital François Mitterrand, Dijon
  - Privé - Cac - Centre Georges-Francois Leclerc, Dijon
  - Privé - Polyclinique de Blois - 3Eme Etage, La Chaussée-Saint-Victor
  - Ch - Chd Vendée, La Roche-sur-Yon
  - CH - GROUPE HOSPITALIER DE La Rochelle RE AUNIS, La Rochelle
  - Privé - Hôpital Franco Britannique, Levallois-Perret
  - Privé - Clinique Du Bois, Lille
  - Chu - Centre Hospitalier Dupuytren, Limoges
  - Ch - Chbs - Hôpital Du Scorff, Lorient
  - Privé - Hôpital Jean Mermoz, Lyon
  - Privé - Hôpital Saint Joseph, Marseille
  - Privé - Hôpital Europeen, Marseille
  - Chu - Hôpital La Timone, Marseille
  - Privé - Haliodx, Marseille
  - Ch - Ghi - Groupe Hospitalier de L'Est Francilien - Site de Meaux, Meaux
  - Ch - Hôpital Layné, Mont-de-Marsan
  - Privé - Centre Azureen de Cancerologie, Mougins
  - Privé - Hôpital Prive Arnault Tzanck, Mougins
  - Privé - Polyclinique de Gentilly, Nancy
  - Chu - Hôpital Carémeau, Nîmes
  - Privé - Institut Mutualiste Montsouris, Paris
  - Chu - Hôpital Europeen Georges Pompidou, Paris
  - Privé - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Chu - Hôpital Saint Antoine, Paris
  - Chu - Hôpital Saint-Louis, Paris
  - Ch - Centre Hospitalier de Pau, Pau
  - Ch - Centre Hospitalier Saint-Jean, Perpignan
  - Chu - Hôpital Haut Lévêque, Pessac
  - Privé - Polyclinique Francheville, Périgueux
  - Chu Lyon Sud - Pierre Benite, Pierre-Bénite
  - Privé - Centre Cario Hpca, Plérin
  - Chu - Centre Hospitalier Universitaire de Poitiers - La Miletrie, Poitiers
  - Ch - Chic de Quimper, Quimper
  - Chu - Centre Hospitalier Universitaire Robert Debre, Reims
  - Privé - Cac - Institut Jean Godinot, Reims
  - Chu - Centre Hospitalier Universitaire Pontchaillou, Rennes
  - Ch - Hôpital Drome Nord, Romans-sur-Isère
  - Privé - Clinique Saint-Grégoire, Saint-Grégoire
  - Privé - Cac - Ico - Site René Gauducheau, Saint-Herblain
  - Chu - Centre Hospitalier Universitaire de Saint Etienne - Hôpital Nord - Service Hge, Saint-Priest-en-Jarez
  - Privé - Polyclinique Saint-Claude, Saint-Quentin
  - Privé - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Ch - Centre Hospitalier de Saint-Malo, St-Malo
  - Privé - Clinique Sainte Anne, Strasbourg
  - Privé - Cac - Paul Strauss / Institut de Cancérologie de Strasbourg Europe, Strasbourg
  - Chu - Hôpital Foch, Suresnes
  - Privé - Polyclinique de L'Ormeau, Tarbes
  - Ch - Hôpital Sainte Musse, Toulon
  - Chu - Hôpital Trousseau, Tours
  - Ch - Centre Hospitalier de Valenciennes, Valenciennes
  - Privé - Cac - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Chu - Hôpital Bradois, Vandœuvre-lès-Nancy
  - Chu - Hôpital Paul Brousse, Villejuif
  - Privé - Cac - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbonnel F, Soularue E, Coutzac C, Chaput N, Mateus C, Lepage P, Robert C. Inflammatory bowel disease and cancer response due to anti-CTLA-4: is it in the flora? Semin Immunopathol. 2017 Apr;39(3):327-331. doi: 10.1007/s00281-016-0613-x. Epub 2017 Jan 16. PMID 28093620
- [Background] Caulet M, Lecomte T, Bouche O, Rollin J, Gouilleux-Gruart V, Azzopardi N, Leger J, Borg C, Douillard JY, Manfredi S, Smith D, Capitain O, Ferru A, Moussata D, Terrebone E, Paintaud G, Ternant D. Bevacizumab Pharmacokinetics Influence Overall and Progression-Free Survival in Metastatic Colorectal Cancer Patients. Clin Pharmacokinet. 2016 Nov;55(11):1381-1394. doi: 10.1007/s40262-016-0406-3. PMID 27312193
- [Background] Diaz LA Jr, Williams RT, Wu J, Kinde I, Hecht JR, Berlin J, Allen B, Bozic I, Reiter JG, Nowak MA, Kinzler KW, Oliner KS, Vogelstein B. The molecular evolution of acquired resistance to targeted EGFR blockade in colorectal cancers. Nature. 2012 Jun 28;486(7404):537-40. doi: 10.1038/nature11219. PMID 22722843
- [Background] Fridman WH, Pages F, Sautes-Fridman C, Galon J. The immune contexture in human tumours: impact on clinical outcome. Nat Rev Cancer. 2012 Mar 15;12(4):298-306. doi: 10.1038/nrc3245. PMID 22419253
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Gordon MS, Margolin K, Talpaz M, Sledge GW Jr, Holmgren E, Benjamin R, Stalter S, Shak S, Adelman D. Phase I safety and pharmacokinetic study of recombinant human anti-vascular endothelial growth factor in patients with advanced cancer. J Clin Oncol. 2001 Feb 1;19(3):843-50. doi: 10.1200/JCO.2001.19.3.843. PMID 11157038
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821
- [Background] Kamphorst AO, Wieland A, Nasti T, Yang S, Zhang R, Barber DL, Konieczny BT, Daugherty CZ, Koenig L, Yu K, Sica GL, Sharpe AH, Freeman GJ, Blazar BR, Turka LA, Owonikoko TK, Pillai RN, Ramalingam SS, Araki K, Ahmed R. Rescue of exhausted CD8 T cells by PD-1-targeted therapies is CD28-dependent. Science. 2017 Mar 31;355(6332):1423-1427. doi: 10.1126/science.aaf0683. Epub 2017 Mar 9. PMID 28280249
- [Background] Lamas B, Richard ML, Leducq V, Pham HP, Michel ML, Da Costa G, Bridonneau C, Jegou S, Hoffmann TW, Natividad JM, Brot L, Taleb S, Couturier-Maillard A, Nion-Larmurier I, Merabtene F, Seksik P, Bourrier A, Cosnes J, Ryffel B, Beaugerie L, Launay JM, Langella P, Xavier RJ, Sokol H. CARD9 impacts colitis by altering gut microbiota metabolism of tryptophan into aryl hydrocarbon receptor ligands. Nat Med. 2016 Jun;22(6):598-605. doi: 10.1038/nm.4102. Epub 2016 May 9. PMID 27158904
- [Background] Misale S, Yaeger R, Hobor S, Scala E, Janakiraman M, Liska D, Valtorta E, Schiavo R, Buscarino M, Siravegna G, Bencardino K, Cercek A, Chen CT, Veronese S, Zanon C, Sartore-Bianchi A, Gambacorta M, Gallicchio M, Vakiani E, Boscaro V, Medico E, Weiser M, Siena S, Di Nicolantonio F, Solit D, Bardelli A. Emergence of KRAS mutations and acquired resistance to anti-EGFR therapy in colorectal cancer. Nature. 2012 Jun 28;486(7404):532-6. doi: 10.1038/nature11156. PMID 22722830
- [Background] Pauken KE, Wherry EJ. Overcoming T cell exhaustion in infection and cancer. Trends Immunol. 2015 Apr;36(4):265-76. doi: 10.1016/j.it.2015.02.008. Epub 2015 Mar 18. PMID 25797516
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Sokol H, Leducq V, Aschard H, Pham HP, Jegou S, Landman C, Cohen D, Liguori G, Bourrier A, Nion-Larmurier I, Cosnes J, Seksik P, Langella P, Skurnik D, Richard ML, Beaugerie L. Fungal microbiota dysbiosis in IBD. Gut. 2017 Jun;66(6):1039-1048. doi: 10.1136/gutjnl-2015-310746. Epub 2016 Feb 3. PMID 26843508
- [Background] Stroun M, Lyautey J, Lederrey C, Olson-Sand A, Anker P. About the possible origin and mechanism of circulating DNA apoptosis and active DNA release. Clin Chim Acta. 2001 Nov;313(1-2):139-42. doi: 10.1016/s0009-8981(01)00665-9. PMID 11694251
- [Background] Thierry AR, Mouliere F, El Messaoudi S, Mollevi C, Lopez-Crapez E, Rolet F, Gillet B, Gongora C, Dechelotte P, Robert B, Del Rio M, Lamy PJ, Bibeau F, Nouaille M, Loriot V, Jarrousse AS, Molina F, Mathonnet M, Pezet D, Ychou M. Clinical validation of the detection of KRAS and BRAF mutations from circulating tumor DNA. Nat Med. 2014 Apr;20(4):430-5. doi: 10.1038/nm.3511. Epub 2014 Mar 23. PMID 24658074
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Vogelstein B, Papadopoulos N, Velculescu VE, Zhou S, Diaz LA Jr, Kinzler KW. Cancer genome landscapes. Science. 2013 Mar 29;339(6127):1546-58. doi: 10.1126/science.1235122. PMID 23539594